CLINICAL TRIAL: NCT06391632
Title: Construction of a Prediction Model for Severe Cardiovascular and Cerebrovascular Complications in Elderly Patients After Elective Non-cardiac Surgery: a Prospective Cohort Study
Brief Title: Construction of a Prediction Model for MACCE in Elderly Patients After Elective Non-cardiac Surgery
Status: Recruiting | Type: Observational
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ZB009
Record Dates: First submitted 2024-04-07; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-03

CONDITIONS: Major Adverse Cardiac Events; Cerebrovascular Accident; Postoperative Complications; Models
Keywords: Elderly patients; Elective non-cardiac surgery; MACCEs; Postoperative Complications; Selective Operation; predictive model
MeSH Terms: conditions — Cardiovascular Diseases; Stroke; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- positive event group: The following complications occur within 3-7 days after surgery：
  1. all-cause death;
  2. non-fatal myocardial infarction/angina pectoris (new or recurring);
  3. non-fatal heart failure (new onset or recurrence);
  4. non-fatal cerebral infarction (new or reappeared);
  5. new or recurrent malignant arrhythmias (ventricular tachycardia/ventricular fibrillation, atrial flutter/atrial fibrillation, hemodynamically unstable second/third degree atrioventricular block);
  Interventions: Diagnostic Test: Revised Cardiac Risk Index
- negative event group: The following complications did not occur within 3-7 days after surgery：
  1. all-cause death;
  2. non-fatal myocardial infarction/angina pectoris (new or recurring);
  3. non-fatal heart failure (new onset or recurrence);
  4. non-fatal cerebral infarction (new or reappeared);
  5. new or recurrent malignant arrhythmias (ventricular tachycardia/ventricular fibrillation, atrial flutter/atrial fibrillation, hemodynamically unstable second/third degree atrioventricular block);
  Interventions: Diagnostic Test: Revised Cardiac Risk Index

INTERVENTIONS:
Diagnostic Test: Revised Cardiac Risk Index — The Revised Cardiac Risk Index (RCRI) attempts to estimate the likelihood of cardiac complications during hospitalization in patients undergoing noncardiac surgery.The Frailty Index is a commonly used tool in clinical practice to assess the degree of frailty in patients.The Quality of Recovery-15 scale (QoR-15) is an easy-to-use score for assessing the quality of post-operative recovery.
  Other Names: Frailty index scale; The Quality of Recovery-15 scale

SUMMARY:
Severe cardiovascular and cerebrovascular complications, including cardiac death, non-fatal angina/myocardial infarction, non-fatal heart failure, stroke, severe arrhythmia, etc., are one of the main types of postoperative complications in elderly patients, and are also the main causes of perioperative death in elderly patients. With the aging population and the large proportion of elderly patients undergoing non-cardiac surgery, it is increasingly important to establish a prediction model for postoperative severe cardiovascular and cerebrovascular events in elderly patients undergoing noncardiac surgery.

DETAILED DESCRIPTION:
This project intends to use a multi-center, prospective cohort study method to include about 3000 elderly patients over 65 years old who are planning to undergo non-cardiac surgery, collect relevant data before, during and after surgery, observe the occurrence of serious cardiovascular and cerebrovascular complications in the perioperative period, establish a "MACCE risk prediction model for elderly patients after elective non-cardiac surgery", and verify its effectiveness and reliability. The results of this study will help to improve the predictive ability of postoperative complications of severe cardiovascular and cerebrovascular events in elderly patients undergoing elective non-cardiac surgery, which is conducive to early risk assessment, risk classification, strengthening perioperative patient management, reducing the incidence of postoperative MACCE, and improving the prognosis of elderly patients.

ELIGIBILITY:
Inclusion Criteria:

* The subjects were patients with elective non-cardiac surgery;
* Older than 65 years;
* Patients signed informed consent.

Exclusion Criteria:

* The anesthesia should be received in any of the following ways: local anesthesia;
* local anesthesia enhancement, and simple nerve block anesthesia;
* Patients who are scheduled to undergo day surgery;
* Expected operation time <1 hour for patients;
* Patients who are expected to stay in hospital for less than 3 days after surgery;
* Patients who refuse to enroll.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients over 65 years of age undergoing elective non-cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiac and Cerebrovascular event（MACCE）occurred in elderly patients after elective non-cardiac surgery | Within 3-7 days after surgery
  1. all-cause death;
  2. non-fatal myocardial infarction/angina pectoris (new or recurring);
  3. non-fatal heart failure (new onset or recurrence);
  4. non-fatal cerebral infarction (new or reappeared);
  5. new or recurrent malignant arrhythmias (ventricular tachycardia/ventricular fibrillation, atrial flutter/atrial fibrillation, hemodynamically unstable second/third degree atrioventricular block);

SECONDARY OUTCOMES:
The Postoperative Quality of Recovery-15 scale (QoR-15) | Postoperative day 1 and postoperative day 3
  The Postoperative Quality of Recovery-15 scale (QoR-15) on the 1st and 3rd postoperative days.The Postoperative Quality of Recovery-15 scale (QoR-15) on the 1st and 3rd postoperative days. The score ranges from 0 to 150, with higher scores indicating better postoperative recovery.
Other complications that occurred during postoperative hospitalization | Until three months after surgery
  Respiratory complications, lower extremity venous thrombosis/pulmonary embolism, renal failure, surgical site infection

CONTACTS AND LOCATIONS:
Overall Officials: Huan Zhang, PhD, Principal Investigator — Beijing Tsinghua Changgeng Hospital
Locations (1):
- Beijing Tsinghua Chang Gung Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided